CLINICAL TRIAL: NCT02706613
Title: A Randomised Controlled Research Study Comparing Online Pulmonary Rehabilitation 'myPR' Versus Conventional Pulmonary Rehabilitation for Patients With COPD
Brief Title: Comparing Online Pulmonary Rehabilitation 'myPR' Versus Conventional Pulmonary Rehabilitation for Patients With COPD
Acronym: TROOPeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: my mhealth Ltd (Industry)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHT/2015/069
Record Dates: First submitted 2015-07-30; First posted 2016-03-11 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Face to Face Pulmonary Rehabilitaton (Other): 6 week incremental pulmonary rehabilitation (PR) programme. Participants will attend 12 sessions over the 6 week period. The components of the PR programme will include an exercise programme. Education sessions will also be provided and include anatomy of the lungs and what is COPD, anxiety and depression, self management, managing breathlessness, medications and treatments, managing exacerbations of COPD and chest infections, clearing sputum and the Active Cycle of Breathing Technique, nutrition, pacing, smoking cessation. Participants on the face to face arm will also be instructed to carry out the pulmonary rehabilitation exercises an additional three times a week at home.
  Interventions: Behavioral: Face to Face Pulmonary Rehabilitaton
- Online Pulmonary Rehabilitation (Active Comparator): Those randomised to receive the online programme will be given log-in details and a password, and instructions to begin the 6 week programme at home. The online programme mirrors the conventional face-to-face PR programme and the exercise and educational components are given by means of instructional videos. Participants will be instructed to exercise five times a week. Participants in the online arm will receive during the PR course telephone contact to record any adverse or serious adverse events.
  Interventions: Behavioral: Online Pulmonary Rehab

INTERVENTIONS:
Behavioral: Face to Face Pulmonary Rehabilitaton — 6 week face to face, incremental exercise and education programme for people with COPD
  Arms: Face to Face Pulmonary Rehabilitaton
Behavioral: Online Pulmonary Rehab — 6 week online, incremental exercise and education programme for people with COPD
  Arms: Online Pulmonary Rehabilitation

SUMMARY:
Over time, patients with COPD (Chronic Obstructive Pulmonary Disease) develop progressive symptoms of breathlessness, which can limit day-to-day activities and tolerance to exercise. Pulmonary Rehabilitation (PR) is an established intervention in the management of COPD and is a structured programme of exercise training and education. Pulmonary Rehabilitation encourages and enables patients to improve their exercise capacity incrementally over the course of a six-week programme. An established evidence base has placed PR at the centre of interventions for COPD and its provision is mandated by NICE as a key pillar of integrated care.

Currently, the provision of PR in the NHS is limited to group sessions run over an established protocol of 6 weeks. Whilst this has been demonstrated to improve exercise capacity, access to PR classes can be problematic for some patients. Also, staff and facility resources limit delivering the programme at scale. An online PR programme developed by my mhealth known as 'myPR', in consultation with patients and physiotherapy experts, offers an alternative provision of this important intervention.

The study aims to compare this online PR programme to conventional face-to-face PR as currently delivered by the NHS. The study aims to recruit 106 patients referred for PR from Portsmouth Hospital and local Participant Identification Centres.They will then be assessed for suitability onto PR, consented and randomised onto an arm of the study. 36 will undertake a conventional PR programme as reflected in the NHS, and 70 the online PR programme known as 'myPR'. Pre and post programme measurements including walking distance and quality of life questionnaires will then be compared between each arm of the trial, to ensure that the online PR is not inferior to the conventional face-to-face PR.

DETAILED DESCRIPTION:
Everyone with Chronic Obstructive Pulmonary Disease (COPD) who is able to exercise should be offered pulmonary rehabilitation (PR). Participants will be invited to take part in the study after being referred for PR by members of Queen Alexandra Hospital (QAH), Portsmouth Hospitals NHS Trust clinical team. They will be given a PIS for the patient to contact the study team to arrange an appointment, or alternatively if verbal consent is obtained the research team will contact the patient to arrange an assessment appointment. Potential participants will also be identified from databases from selected GP who meet the protocol inclusion and exclusion criteria. These potential participants will be sent a study participation invitation letter and asked to contact the respiratory research team at QAH to arrange an assessment appointment.

If a participant decides they would like to take part and contacts the respiratory research team or have been contacted by the team, an initial appointment will be arranged. This will take part at the participants home, GP surgery or Queen Alexandra Hospital depending on the patients choice. After obtaining consent, suitability for inclusion onto pulmonary rehabilitation will be assessed. A full medical history (including confirmation of diagnosis, COPD severity, smoking history, medications and current activity) along with blood pressure will be taken to assess for any exclusion criteria. The timed "Up and Go" Test will also be performed to assess safety of mobility and exercising. This is to ensure it is safe for the participant to exercise independently. If a participant does not meet the inclusion criteria, they will be referred back to their GP with the reason they were not suitable for PR. It is explained to the participant that they can withdraw from the study at any point and that this will not affect their care. If a participant decides they do not wish to be included onto the study they will be referred to the conventional NHS PR programme. If a participant is suitable for PR and is willing to participate, further screening is undertaken. This can take place immediately if this initial appointment is carried out at QAH, or a further appointment will be arranged at QAH will be arranged.

The next stage of the assessment (this may be a further appointment (visit 2) if the initial assessment was not carried out a QAH) will take place at Queen Alexandra Hospital where the space is available to carry out the assessments. Transport can be provided to this venue if required. Consent will first be obtained and participants will then complete the first of two walking test for 6 minutes to measure how far they can walk, known as the six-minute walking test . Oxygen levels will be measured using a probe that fits on the finger and if significant oxygen desaturation is noted, the participant will be withdrawn from the study and referred onto the local oxygen assessment centre. The participant will be asked to fill out four health- related questionnaires and they will then repeat the six minute walking test and the best of the two tests will be recorded.

If the participant is suitable to undertake a PR programme they will then be randomised to either receive the online PR 'my PR', or the conventional face-to-face PR. Randomisation will be undertaken by an online randomisation system hosted by my mhealth.

Participants randomised to receive the conventional PR will be given 12 visit dates (twice a week for six weeks) at the PR venue where the face-to-face sessions will take place. This attendance length and frequency is standard for PR. The components of the PR programme will include an exercise programme, including a warm-up and cool- down programme. Education sessions will also be provided and includes anatomy of the lungs and what is COPD, anxiety and depression, claiming benefits, self management, managing breathlessness, medications and treatments, managing exacerbations of COPD and chest infections, clearing sputum and the Active Cycle of Breathing Technique, nutrition, pacing, smoking cessation and advice on travel with COPD. Participants on the face to face arm will also be instructed to carry out the pulmonary rehabilitation exercises an additional three times a week at home. An exercise leaflet used in the PR classes will be given to be filled out at home.

Those randomised to receive the online programme will be loaned a computer/tablet for the six-week duration, given log-in details and a password, and instructions to begin the programme at home. A further visit to these participants home may need to be arranged to ensure that the Internet connection is suitable. If the internet connection is unsuitable, the participant will be withdrawn from the study and referred to the NHS PR. The online programme mirrors the conventional face-to-face PR programme and the exercise and educational components are given by means of instructional videos. Participants will be instructed to exercise five times a week. Participants in the online arm will receive during the PR course telephone contact to record any adverse or serious adverse events. They will be contacted twice during the first 2 weeks, then weekly for the remaining 5 weeks.

After completing the 6- week online PR or the 6- week conventional PR, participants will have their final visit arranged which will take place at the Queen Alexandra Hospital. The pre-PR measurements including the two 6-minute walking tests and quality of life questionnaires will be repeated, and results collected. These measurements will be statistically analysed for comparison between the two arms of the study to ensure the online PR is not inferior to face-to-face PR.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to complete all study procedures and give written informed consent.
2. A diagnosis of COPD defined as per the NICE COPD guidelines with an MRC score of 2 or greater or appropriately symptomatic patients.
3. Male or female volunteers aged 40+ with a diagnosis of COPD referred for pulmonary rehabilitation
4. Access to the internet and ability to operate a web platform

Exclusion Criteria:

1. Patients who have had an exacerbation requiring additional antibiotics and/or an additional course of steroids within 2 weeks prior to commencing the study.
2. Patients who have already undertaken a pulmonary rehabilitation programme within the last 6 months
3. Patients who have another respiratory disease as their main complaint, such as asthma, bronchiectasis, lung cancer, tuberculosis or any other significant respiratory disease.
4. Uncontrolled hypertension
5. Unstable cardiovascular disease that would make pulmonary rehabilitation exercise unsafe or prevent programme participation
6. Patients who are unable to walk or whose ability to walk safely and independently is significantly impaired due to non-respiratory related conditions and/or cognitive impairment
7. Patients who are unable to read, or use an internet enabled device or do not have access to the internet at home
8. A timed 'Up and Go' test greater than 14 seconds

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Distance | 6 weeks
  The 6- minute walking distance (6MWD) is assessed by carrying out the 6 Minute Walk Test (6MWT).The aim of the 6MWT is to measure walking endurance and distance over a 30m course. The patient is asked to walk as far as possible along a designated course, at a self-regulated rate for 6 minutes. Within this time they can stop and rest as needed. The patient's final walking distance is recorded (6MWD).
COPD Assesment Tool (CAT) | 6 weeks
  This is a validated symptom-scoring questionnaire used in COPD studies. The CAT questionnaire contains 8 questions and provides a reliable measure of the impact of COPD on health status. The higher the CAT score the greater the impact on health staus.

SECONDARY OUTCOMES:
St Georges Respiratory Questionnaire | 6 weeks
  This is a validated symptom-scoring questionnaire used in COPD studies. The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction. Scores are calculated for three domains Symptoms, Activity and Impacts (Psycho-social).
Hospital Anxiety and Depression scale | 6 weeks
  This was developed to determine the levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen-item scale. Seven of the items relate to anxiety and seven relate to depression.11 If a participant scores higher than 8/21 on either the anxiety or depression scale, a letter will be sent to their GP informing them of their patients abnormal score so that a consultation can be arranged and treatment be provided as required.
Modified Medical Research Council Dyspnoea scale | 6 weeks
  The MRC breathlessness scale comprises five statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). It is self-administered by asking subjects to choose a phrase that best describes their condition, e.g. 'I only get breathless with strenuous exertion' (Grade 1) or 'I am too breathless to leave the house' (Grade 5). The score is the number that best fits the patient's level of activity. All the questions relate to everyday activities and are easily understood by patients
Safety | 6 weeks
  Safety will be evaluated from reported adverse and serious adverse evenets reported by the patients during the 6 week intervention
Adherence | 6 week
  A register of attendance will be maintained in the face to face arm. In the online arm the number of days accessing the online programme will be recorded
Usability of online platform | 6 weeks
  This qualitative information will be obtained by using a feedback form

CONTACTS AND LOCATIONS:
Overall Officials: Ben Green, Dr, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospital NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Result] Sewell L, Singh SJ, Williams JE, Collier R, Morgan MD. [Can individualized rehabilitation improve functional independence in elderly patients with COPD?]. Rev Port Pneumol. 2005 Nov-Dec;11(6):593-6. No abstract available. Portuguese. PMID 16514719
- [Result] Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM. Regular physical activity reduces hospital admission and mortality in chronic obstructive pulmonary disease: a population based cohort study. Thorax. 2006 Sep;61(9):772-8. doi: 10.1136/thx.2006.060145. Epub 2006 May 31. PMID 16738033
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831
- [Result] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Result] Snaith RP, Zigmond AS. The hospital anxiety and depression scale. Br Med J (Clin Res Ed). 1986 Feb 1;292(6516):344. doi: 10.1136/bmj.292.6516.344. No abstract available. PMID 3080166
- [Result] Redelmeier DA, Bayoumi AM, Goldstein RS, Guyatt GH. Interpreting small differences in functional status: the Six Minute Walk test in chronic lung disease patients. Am J Respir Crit Care Med. 1997 Apr;155(4):1278-82. doi: 10.1164/ajrccm.155.4.9105067.
- [Result] Troosters T, Gosselink R, Decramer M. Six minute walking distance in healthy elderly subjects. Eur Respir J. 1999 Aug;14(2):270-4. doi: 10.1034/j.1399-3003.1999.14b06.x. PMID 10515400
- [Result] Kon SS, Canavan JL, Jones SE, Nolan CM, Clark AL, Dickson MJ, Haselden BM, Polkey MI, Man WD. Minimum clinically important difference for the COPD Assessment Test: a prospective analysis. Lancet Respir Med. 2014 Mar;2(3):195-203. doi: 10.1016/S2213-2600(14)70001-3. Epub 2014 Feb 4. PMID 24621681
- [Result] Cote CG, Casanova C, Marin JM, Lopez MV, Pinto-Plata V, de Oca MM, Dordelly LJ, Nekach H, Celli BR. Validation and comparison of reference equations for the 6-min walk distance test. Eur Respir J. 2008 Mar;31(3):571-8. doi: 10.1183/09031936.00104507. Epub 2007 Nov 7. PMID 17989117
- [Result] Fletcher CM. Standardised questionnaire on respiratory symptoms: a statement prepared and approved by the MRC Committee on the Aetiology of Chronic Bronchitis (MRC breathlessness score). BMJ 1960; 2: 1665.
- [Result] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Result] Mesquita R et al. Timed Up and Go test in COPD: Changes over time, validity and responsiveness to pulmonary rehabilitation. ERJ September1, 2014 vol 44 suppl 58 P3037
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- See also: NICE COPD Guidelines — https://www.nice.org.uk/guidance/cg101